CLINICAL TRIAL: NCT02396095
Title: Live Birthrate Following Oocyte Cryopreservation
Brief Title: Oocyte Cryopreservation Study (Egg Banking)
Status: Terminated | Type: Observational
Why Stopped: American Society of Reproductive Medicine guidelines, October 2012.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Clarisa Gracia, Clarisa R. Gracia, MD, MSCE, University of Pennsylvania
Other Study IDs: 808392
Record Dates: First submitted 2015-03-17; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Cancer
Keywords: female; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — oocytes
Oversight: Data Monitoring Committee: No

SUMMARY:
Women of reproductive age who seek to freeze eggs for future pregnancy attempts may be eligible to participate in a study investigating pregnancies that result from frozen eggs.

DETAILED DESCRIPTION:
Participants follow standard fertility protocols to stimulate the growth of multiple egg follicles. When the egg follicles are mature, the eggs will be removed under sedation, examined by an embryologist under a microscope and the mature eggs will be immediately frozen and kept frozen in tanks at Penn Fertility Care using the same methods of labeling and quality assurance currently in place for frozen embryos.

Eggs will be thawed in the future when the participant wishes to attempt pregnancy and fertilized by standard methods used during In Vitro Fertilization (IVF). Resulting embryos will be placed into the uterus by a procedure that will require approximately 15-30 minutes. The number of embryos to be transferred will be dictated by standard clinical practice. After embryo transfer, subjects will return for serum pregnancy tests at 14 days after the embryo transfer. For those who are not pregnant, there will be no further participation in the study. For those who do achieve pregnancy, trans-vaginal ultrasound will be performed at approximately 6 weeks gestation and weekly thereafter until 8 weeks gestation at which time, they will be referred to their general obstetrician for prenatal care. Participants will be asked to provide the study team with information about birthweight, height, length, gestational age at delivery, complications at delivery, and infant number. This information is routinely collected from patients undergoing conventional IVF in order to maintain quality assurance as recommended by the American Society of Reproductive Medicine. Information will also be collected from the participant's medical records including physical characteristics, medical and fertility history, semen analysis of the partner if appropriate, egg stimulation characteristics including medications, days of stimulation, number of egg follicles, number of mature and immature eggs retrieved, number of eggs frozen, number of eggs thawed, number of embryos, disposition of embryos, pregnancy test results, number of pregnancies that survived the first 12 weeks and prenatal screening tests.

ELIGIBILITY:
Inclusion Criteria:

* age between 15 and 45
* desire oocyte cryopreservation or use of cryopreserved oocytes for the purposes of achieving pregnancy
* willingness to participate in study and provide informed consent

Exclusion Criteria:

* day 3 FSH over 20 mIU/ml, or Day 3 E2 over 100pg/ml
* ovarian cyst greater than 14mm at baseline ultrasound
* uncontrolled medical illness such as diabetes, hypertension, or cardiovascular disease
* current pregnancy

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Penn Fertility Care
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Live birthrate following transfer of embryos created from frozen eggs | 10 years
  Live birthrate following transfer of embryos created from frozen eggs in the setting of: Autologous oocyte cryopreservation in women without cancer vs.autologous oocyte cryopreservation in women with cancer.

SECONDARY OUTCOMES:
Oocyte survival rates | 10 years
  The number of oocytes surviving cryopreservation, storage, and thaw will be evaluated.

OTHER OUTCOMES:
Fertilization rates | 10 years
  Fertilization rates in each cohort will be compared.
Perinatal outcomes | 10 years
  Perinatal outcomes in each cohort will be evaluated including birth weight and gestational age at delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa R Gracia, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Reproductive Research Unit, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Oncofertility — http://www.uphs.upenn.edu/obgyn/clinical-trials/